CLINICAL TRIAL: NCT03817190
Title: A Randomised, Double-blind, Placebo-controlled, Study to Assess the Efficacy and Safety of Orally Administered DS107 in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Safety of Orally Administered DS107 in Adult Patients With Moderate to Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on Interim Analysis results
Sponsor: DS Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS107G-05-AD3
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Results first posted 2022-05-06 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — 8,11,14-Eicosatrienoic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2g Oral DS107 (Experimental): 2g DS107 (4 DS107 capsules) administered once-daily for 16 weeks
  Interventions: Drug: DS107
- Placebo (Placebo Comparator): Placebo (4 placebo capsules) orally administered once-daily for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS107 — DS107 Capsule
  Other Names: DS107 500mg DGLA Capsules/DS107 500mg Placebo Capsules
  Arms: 2g Oral DS107
Drug: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the efficacy and safety of orally administered DS107 (2g) versus placebo in the treatment of moderate to severe Atopic Dermatitis (AD).

Oral DS107/Placebo capsules will be administered for 16 weeks. The study will enrol approximately 220 subjects.

DETAILED DESCRIPTION:
This study involves a comparison of 2g DS107 with placebo, administered orally once daily for a total of 16 weeks. Patients will be randomized to one of the two treatment arms in a 1:1 ratio.

The primary endpoint will be the vIGA (Validated Investigator's Global Assessment) and EASI (Eczema Area and Severity Index). Other endpoints include vIGA, EASI, SCORAD, BSA (Body Surface Area) and NRS (Numeric Rating Scale).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clinically confirmed diagnosis of active AD according to the American Academy of Dermatology Consensus Criteria that had been present for at least 6 months before the screening visit.
2. Patients with moderate to severe AD at baseline as defined by a Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-ADTM) score of 3 Or 4 at baseline.
3. Patients with an Eczema Area and Severity Index (EASI) score of ≥16 at screening and baseline.
4. Patients with AD covering a minimum 10% of the Body Surface Area (BSA) at baseline.
5. Patients with a worst itch Numeric Rating Scale (NRS) score in a day of ≥4 (on 11-point NRS) at the screening and baseline visits.
6. Patients whose pre-study clinical laboratory findings did not interfere with their participation in the study, in the opinion of the investigator.
7. Patients who were able and willing to stop all current treatments for AD throughout the study (except for allowed emollients).
8. Patients who were on a stable dose of a bland emollient for at least 7 days prior to baseline.
9. Male or female patients aged 18 years and older on the day of signing the informed consent form (ICF).
10. Female patients and male patients with female partners of child bearing potential had to use highly effective birth control methods or have a sterilised partner for the duration of the study.
11. Recent history (within 6 months before the screening visit) of inadequate response to treatment with topical medications or for whom topical treatments were otherwise medically inadvisable (e.g. because of important side effects or safety risks).
12. Patients who were able to communicate well with the investigator, to understand and comply with the requirements of the study, and understand and sign the written informed consent prior to initiation of any study specific activities or procedures.

Exclusion Criteria:

1. Patients with other skin conditions that might interfere with AD diagnosis and/or evaluation (such as psoriasis or current active viral, bacterial and fungal topical skin infections) as assessed by the investigator.
2. Patients who had used systemic treatments that could affect AD less than 4 weeks prior to Baseline Visit (Day 0), e.g. retinoids, methotrexate, cyclosporine, hydroxycarbamide (hydroxyurea), azathioprine and oral/injectable corticosteroids.

   Intranasal corticosteroids and inhaled corticosteroids for stable medical conditions were allowed.
3. Patients with previous exposure to DS107.
4. Patients who had used any topical medicated treatment for AD (except for emollients) two weeks prior to start of treatment/Baseline (Day 0) including but not limited to, topical corticosteroids, calcineurin inhibitors, tars, bleach, antimicrobials and bleach baths.
5. Patients who used emollients containing urea, ceramides or hyaluronic acid less than 12 weeks prior to Baseline (Day 0).
6. Patients who have had excessive sun exposure, have used tanning booths or other ultraviolet (UV) light sources four weeks prior to Baseline (Day 0) and/or were planning a trip to a sunny climate or to use tanning booths or other UV sources between screening and follow-up visits.
7. Patients who had a history of hypersensitivity to any substance in DS107 or placebo capsules.
8. Patients who had a history of hypersensitivity to soy beans or soy lecithin.
9. Patients who had a white cell count or differential white cell count outside of the normal reference range at screening.
10. Patients who had any clinically significant controlled or uncontrolled medical condition or laboratory abnormality that would, in the opinion of the investigator, put the patient at undue risk or interfere with interpretation of study results.
11. Patients who had a clinically significant impairment of renal or hepatic function.
12. Patients with significant uncontrolled cardiovascular, neurologic, malignant, psychiatric, respiratory or hypertensive disease, as well as uncontrolled diabetes and fluoride arthritis or any other illness that, in the opinion of the investigator, was likely to interfere with completion of the study.
13. Patients with active infectious diseases (e.g. hepatitis B, hepatitis C or advanced disease secondary to infection with human immunodeficiency virus).
14. Patients with a history of clinically significant drug or alcohol abuse in the opinion of the investigator in the last year prior to Baseline (Day 0).
15. Patients who had participated in any other clinical study with an investigational drug within 3 months before the first day of administration of study treatment.
16. Patients who have had treatment with biologics as follows:

    Any cell-depleting agents including but not limited to rituximab: within 6 months before the screening visit, or until lymphocyte count returned to normal, whichever was longer. b. Other biologics influencing cell proliferation: within 6 months before the screening visit. c. Dupilumab or other monoclonal antibodies within 5 half-lives (if known) or 16 weeks prior to baseline visit, whichever was longer.
17. Patients who were pregnant, planning pregnancy, breastfeeding and/or were unwilling to use adequate contraception (as specified in Inclusion Criterion 10) during the trial.
18. Patients, in the opinion of the investigator, not suitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Weissbach, MD, Study Chair — DS Biopharma
Locations (50):
- United States (26):
  - DS Investigational Site 524, Birmingham, Alabama
  - DS Investigational Site 528, Huntington Beach, California
  - DS Investigational Site 502, Los Angeles, California
  - DS Investigational Site 504, San Diego, California
  - DS Investigational Site 505, San Diego, California
  - DS Investigational Site 516, Santa Ana, California
  - DS Investigational Site 501, Santa Monica, California
  - DS Investigational Site 517, Washington D.C., District of Columbia
  - DS Investigational Site 527, Doral, Florida
  - DS Investigational Site 510, Sunrise, Florida
  - DS Investigational Site 512, Columbus, Georgia
  - DS Investigational Site 514, Skokie, Illinois
  - DS Investigational Site 513, Louisville, Kentucky
  - DS Investigational Site 519, Troy, Michigan
  - DS Investigational Site 511, Raleigh, North Carolina
  - DS Investigational Site 526, Grants Pass, Oregon
  - DS Investigational Site 521, Medford, Oregon
  - DS Investigational Site 525, Philadelphia, Pennsylvania
  - DS Investigational Site 509, Arlington, Texas
  - DS Investigational Site 506, Austin, Texas
  - DS Investigational Site 508, Cypress, Texas
  - DS Investigational Site 507, San Antonio, Texas
  - DS Investigative Site 529, Orem, Utah
  - DS Investigative Site 530, Salt Lake City, Utah
  - DS Investigational Site 523, Richmond, Virginia
  - DS Investigational Site 518, Kenosha, Wisconsin
- DS Investigational Site 101, Graz, Austria
- Germany (12):
  - DS Investigational Site 203, Augsburg
  - DS Investigational Site 202, Berlin
  - DS Investigational Site 208, Berlin
  - DS Investigational Site 204, Dresden
  - DS Investigational Site 206, Essen
  - DS Investigational Site 201, Frankfurt
  - DS Investigational Site 207, Gera
  - DS Investigational Site 211, Leipzig
  - DS Investigational Site 205, Lübeck
  - DS Investigational Site 210, Mainz
  - DS Investigational Site 214, Münster
  - DS Investigational Site 212, Rostock
- Latvia (5):
  - DS Investigational Site 304, Jūrmala
  - DS Investigational Site 301, Riga
  - DS Investigational Site 302, Riga
  - DS Investigational Site 303, Riga
  - DS Investigational Site 305, Riga
- Poland (6):
  - DS Investigational Site 406, Gdansk
  - DS Investigational Site 402, Lodz
  - DS Investigational Site 403, Poznan
  - DS Investigational Site 405, Warsaw
  - DS Investigational Site 407, Warsaw
  - DS Investigational Site 401, Wroclaw

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 219 patients were randomised in a 1:1 ratio.
Groups:
- Placebo: Placebo (4 placebo capsules) orally administered once daily for 16 weeks.
- DS107 2000mg: 2g DS107 (4 DS107 capsules) orally administered once daily for 16 weeks.
Period: Overall Study
Arm/Group | Placebo | DS107 2000mg
Started | 110 | 109
Completed | 50 | 50
Not Completed | 60 | 59
Not completed — Early Termination | 13 | 20
Not completed — Adverse Event | 10 | 17
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Lost to Follow-up | 11 | 7
Not completed — Lack of Efficacy | 7 | 5
Not completed — Investigator Decision | 5 | 1
Not completed — Due to Coronavirus, the patient did not want to continue the study. | 0 | 1
Not completed — Lack of Contact | 1 | 0
Not completed — Due to worsening of atopic dermatitis and use of Con Med, patient was excluded | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Randomised Set consists of all patients who are randomised to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DS107 2000mg | Total
Number analyzed (Participants) | 110 | 109 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.95 (14.90) | 38.83 (15.45) | 38.38 (15.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 55 | 115
  Male | 50 | 54 | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 18 | 35
  White | 90 | 87 | 177
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Body Surface Area Affected [Mean (Standard Deviation); unit: Percentage of body surface area] | 35.95 (17.69) | 35.67 (18.08) | 35.81 (17.85)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving a Validated Investigator Global Assessment Scale for Atopic Dermatitis Score of 0 or 1 and a Decrease of at Least 2 Points in vIGA-ADTM in Treated Population Compared to Placebo Population From Baseline at Week 16.
Description: Proportion of patients achieving a Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-ADTM) score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in vIGA-ADTM in treated population compared to placebo population from Baseline at Week 16 using GLMM.The vIGA-ADTM scale awards a score of 0-4 based on a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease). The scale uses clinical characteristics of erythema, infiltration, papulation and oozing/crusting as scoring guidelines for the overall severity assessment.
Time Frame: 16 Weeks
Population: Full analysis set - consists of all patients who were randomised to the study and received at least one dose of study medication. FAS was the primary analysis population for efficacy endpoints. Analysis was done according to the treatment patients were randomised to.
Measure: Number; unit: Number of participants
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 86 | 92
Number of participants | 15 | 14
Statistical Analysis 1: Comparison: Placebo vs DS107 2000mg; Test type: Superiority; p = 0.6880, GLMM; Proportion of participants = -0.2277, 95% CI 2-sided [-1.0415 to 0.5860]

2. Primary Outcome: Proportion of Patients Achieving EASI-75 in Treated Population Compared to Placebo Population at Week 16.
Description: Proportion of patients achieving EASI-75 (≥75% improvement from Baseline) in treated population compared to placebo population at Week 16 using GLMM.
Time Frame: 16 Weeks
Population: Full analysis set consists of all patients who were randomised to the study, received at least one dose of study medication and whom reached week 16. Analysis was done according to the treatment patients were randomised to.
Measure: Number; unit: participants
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 87 | 93
participants | 30 | 27
Statistical Analysis 1: Comparison: Placebo vs DS107 2000mg; Test type: Superiority; p = 0.4321, GLMM; Proportion of participants = -0.2760, 95% CI 2-sided [-0.9185 to 0.3665]

3. Secondary Outcome: Proportion of Patients Achieving a vIGA-ADTM Score of 0 or 1 and a Decrease of at Least 2 Points in vIGA-ADTM in Treated Population Compared to Placebo Population From Baseline to Week 4, 8, 12, 18 and 20.
Description: Proportion of patients achieving a Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-ADTM) score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in vIGA-ADTM in treated population compared to placebo population from baseline to Week 4, 8, 12, 18 and 20 and the change in proportion of patients from Week 16 to Week 18 and 20.
  The vIGA-ADTM scale awards a score of 0-4 based on a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease). The scale uses clinical characteristics of erythema, infiltration, papulation and oozing/crusting as scoring guidelines for the overall severity assessment.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 18 and Week 20.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 102 | 99
participants
  Baseline to Week 4: number analyzed (Participants) | 83 | 77
  Baseline to Week 4 | 3 | 2
  Baseline to Week 8: number analyzed (Participants) | 63 | 58
  Baseline to Week 8 | 6 | 6
  Baseline to Week 12: number analyzed (Participants) | 49 | 45
  Baseline to Week 12 | 10 | 7
  Baseline to Week 18: number analyzed (Participants) | 55 | 51
  Baseline to Week 18 | 13 | 7
  Baseline to Week 20: number analyzed (Participants) | 49 | 46
  Baseline to Week 20 | 10 | 13
  Week 16 to Week 18: number analyzed (Participants) | 55 | 51
  Week 16 to Week 18 | 1 | 1
  Week 16 to Week 20: number analyzed (Participants) | 49 | 46
  Week 16 to Week 20 | 2 | 1

4. Secondary Outcome: Proportion of Patients Achieving EASI-75 (≥75% Improvement From Baseline) in Treated Population Compared to Placebo Population at Weeks 4, 8, 12, 18 and 20
Description: Proportion of Patients Achieving EASI-75 (≥75% Improvement in Eczema Area and Severity Index from Baseline) in Treated Population Compared to Placebo Population at Weeks 4, 8, 12, 18 and 20 EASI quantifies the severity of a patient's AD based on both lesion severity and the percent of BSA affected. The EASI is a composite score ranging from 0-72 that takes into account the degree of erythema, induration/papulation, excoriation, and lichenification (each scored from 0 to 3 separately, half points are permitted) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 18 and Week 20.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 102 | 99
participants
  Baseline to Week 4 | 8 | 8
  Baseline to Week 8 | 15 | 7
  Baseline to Week 12 | 19 | 10
  Baseline to Week 18 | 21 | 20
  Baseline to Week 20 | 23 | 22

5. Secondary Outcome: Change From Baseline in Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-ADTM) Score in Treated Population Compared to Placebo Population to Weeks 4, 8, 12, 16, 18 and 20.
Description: The Validated Global Investigator Assessment scale for Atopic Dermatitis (vIGA-AD) scale awards a score of 0-4 based on a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease). The scale uses clinical characteristics of erythema, infiltration, papulation and oozing/crusting as scoring guidelines for the overall severity assessment. A decrease in Validated Global Investigator Assessment scale indicates a positive outcome for the participant.
Time Frame: 20 Weeks
Population: FAS consists of all patients who were randomised to the study and received at least one dose of study medication. FAS was the primary analysis population for efficacy endpoints. Analysis was done according to the treatment patients were randomised to.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 102 | 99
Scores on a scale
  Week 4 vs Baseline | 0.7843 [0.4869 to 1.0816] | -0.0454 [-0.4715 to 0.3807]
  Week 8 vs Baseline | 0.3487 [0.03437 to 0.6630] | 0.2577 [-0.1929 to 0.7083]
  Week 12 vs Baseline | 0.1224 [-0.2109 to 0.4558] | 0.3091 [-0.1687 to 0.7870]
  Week 16 vs Baseline | 0.2813 [-0.01342 to 0.5761] | 0.1394 [-0.2781 to 0.5568]
  Week 18 vs Baseline | 0.0862 [-0.2366 to 0.4089] | 0.1283 [-0.3349 to 0.5914]
  Week 18 vs Last Visit ( Week 20) | 0.0689 [-0.2153 to 0.3531] | 0.1024 [-0.3055 to 0.5102]

6. Secondary Outcome: Change From Baseline in EASI in Treated Population Compared to Placebo Population to Weeks 4, 8, 12, 16, 18 and 20.
Description: Change from Baseline in Eczema Area and Severity Index (EASI) in treated population compared to placebo population to Weeks 4, 8, 12, 16, 18 and 20. EASI quantifies the severity of a patient's atopic dermatitis (AD) based on both lesion severity and the percent of body surface area (BSA) affected.
  The EASI is a composite score ranging from 0 (no lesion severity) to 72 (severe lesions) that takes into account the degree of erythema, induration/papulation, excoriation, and lichenification (each scored from 0 to 3 separately, half points are permitted) for each of four body regions, with adjustment for the percent of Body Surface Area (BSA) involved for each body region and for the proportion of the body region to the whole body. The severity of each sign is assessed using a 4-point scale (half points are permitted):
  * 0 = none
  * 1 = mild
  * 2 = moderate
  * 3 = severe A decrease in EASI indicates a positive outcome for the participant.
Time Frame: Week 20
Population: Full analysis set consists of all patients who were randomised to the study and received at least one dose of study medication. FAS was the primary analysis population for efficacy endpoints. Analysis was done according to the treatment patients were randomised to.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 102 | 99
Scores on a scale
  Week 4 vs Basline | 31.4509 [17.6525 to 45.2493] | 3.5453 [-16.1397 to 23.2303]
  Week 8 vs Baseline | 14.4747 [-0.08487 to 29.0342] | 8.8565 [-11.9180 to 29.6310]
  Week 12 vs Baseline | 6.4487 [-8.9305 to 21.8279] | 10.4186 [-11.6294 to 32.4667]
  Week 16 vs Baseline | 18.4269 [4.8107 to 32.0431] | 3.5470 [-15.6720 to 22.7661]
  Week 18 vs Baseline | 4.1677 [-10.7908 to 19.1262] | 3.1252 [-18.2311 to 24.4815]
  Week 18 vs Last Visit (Week 20) | 2.6189 [-53.4435 to 58.6812] | 10.1487 [-70.3673 to 90.6647]

7. Secondary Outcome: Change From Baseline in Worst Itch NRS in Treated Population Compared to Placebo Population to Week 4, 8, 12, 16, 18.
Description: Change from Baseline in worst itch Numeric Rating Scale (NRS) in treated population compared to placebo population to Week 4, 8, 12, 16 and 18. Severity of pruritus related to atopic dermatitis (AD) was self-assessed by patients daily using the NRS. Patients were asked to estimate the intensity of pruritus at its worst over the previous 24 hours. The Pruritus NRS is a single-question assessment tool that was used to assess the patient's worst itch as a result of AD in the previous 24 hours. Patients will score their pruritus due to AD on a scale of 0 - 10, with 0 indicating no itch and 10 indicating the worst itch imaginable. Patients will complete the rating scale daily starting at screening through to the last study visit. A decrease in worst itch NRS indicates a positive outcome for the participant.
Time Frame: Week 18
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 102 | 99
score on a scale
  Week 4 vs Baseline | 1.9916 [1.1339 to 2.8493] | -0.5094 [-1.7037 to 0.6848]
  Week 8 vs Baseline | 1.2897 [0.4072 to 2.1723] | -0.2826 [-1.5060 to 0.9408]
  Week 12 vs Baseline | 0.8685 [-0.05200 to 1.7889] | -0.2133 [-1.4913 to 1.0646]
  Week 16 vs Baseline | 0.2244 [-0.7377 to 1.1865] | 0.0258 [-1.3063 to 1.3579]
  Week 18 vs Baseline | 0.0905 [-0.9063 to 1.0873] | 0.1468 [-1.2412 to 1.5348]

8. Secondary Outcome: Proportion of Patients Achieving a Decrease of at Least 3 Points in Worst Itch NRS in Treated Population Compared to Placebo Population From Baseline to Week 4, 8, 12, 16, 18 and 20.
Description: Proportion of Patients Achieving a Decrease of at Least 3 Points in Worst Itch Numeric Rating Scale (NRS) in Treated Population Compared to Placebo Population From Baseline to Week 4, 8, 12, 16, 18 and 20.
  The Pruritus NRS is a single-question assessment tool that will be used to assess the patient's worst itch as a result of AD in the previous 24 hours. Patients score their pruritus due to AD on a scale of 0 - 10, with 0 (no itch) and 10 (worst itch imaginable). Patients will complete the rating scale daily starting at screening through to the last study visit.
Time Frame: Week 20
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 102 | 99
participants
  Week 4 | 12 | 19
  Week 8 | 18 | 22
  Week 12 | 21 | 21
  Week 16 | 20 | 22
  Week 18 | 17 | 16
  Week 20 | 16 | 16

9. Secondary Outcome: Proportion of Patients Achieving a Decrease of at Least 4 Points in Worst Itch NRS in Treated Population Compared to Placebo Population From Baseline to Week 4, 8, 12, 16, 18 and 20,
Description: Proportion of patients achieving a decrease of at least 4 points in worst itch Numeric Rating Scale (NRS) in treated population compared to placebo population from baseline to Week 4, 8, 12, 16, 18 and 20. Severity of pruritus related to atopic dermatitis (AD) was self-assessed by patients daily using the NRS. Patients were asked to estimate the intensity of pruritus at its worst over the previous 24 hours. The Pruritus NRS is a single-question assessment tool that is used to assess the patient's worst itch as a result of AD in the previous 24 hours. Patients will score their pruritus due to AD on a scale of 0 - 10, with 0 indicating no itch and 10 indicating the worst itch imaginable. Patients completed the rating scale daily starting at screening through to the last study visit. A decrease in worst itch NRS indicates a positive outcome for the participant.
Time Frame: Week 20
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 102 | 99
participants
  Week 4 | 6 | 11
  Week 8 | 12 | 12
  Week 12 | 10 | 13
  Week 16 | 13 | 12
  Week 18 | 12 | 12
  Week 20 | 11 | 10

10. Secondary Outcome: Proportion of Patients Achieving EASI-50 (≥50% Improvement From Baseline) in Treated Population Compared to Placebo Population at Week 4, 8, 12, 16, 18 and 20.
Description: Proportion of Patients Achieving EASI-50 (≥50% Improvement in Eczema Area and Severity Index From Baseline) in Treated Population Compared to Placebo Population at Week 4, 8, 12, 16, 18 and 20.
  The EASI is a composite score ranging from 0-72 that takes into account the degree of erythema, induration/papulation, excoriation, and lichenification (each scored from 0 to 3 separately, half points are permitted) for each of four body regions, with adjustment for the percent of Body Surface Area (BSA) involved for each body region and for the proportion of the body region to the whole body. The severity of each sign is assessed using a 4-point scale (half points are permitted):
  * 0 = none
  * 1 = mild
  * 2 = moderate
  * 3 = severe A decrease in EASI indicates a positive outcome for the participant.
Time Frame: Week 20
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 102 | 99
participants
  Week 4 | 21 | 15
  Week 8 | 31 | 26
  Week 12 | 28 | 23
  Week 16 | 44 | 45
  Week 18 | 29 | 35
  Week 20 | 29 | 33

11. Secondary Outcome: Change From Baseline in the Body Surface Area Affected by AD in Treated Population Compared to Placebo Population to Weeks 4, 8, 12, 16, 18.
Description: Change from Baseline in the Body Surface Area (BSA) affected by AD in treated population compared to placebo population to Weeks 4, 8, 12, 16, 18.
Time Frame: Week 18
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: % Change from Baseline
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 102 | 99
% Change from Baseline
  Week 4 vs Baseline | 10.5575 [5.0467 to 16.0682] | -1.1911 [-9.0736 to 6.6913]
  Week 8 vs Baseline | 7.0087 [1.1680 to 12.8495] | -0.2839 [-8.6398 to 8.0720]
  Week 12 vs Baseline | 4.8296 [-1.3215 to 10.9808] | -1.4232 [-10.2908 to 7.4445]
  Week 16 vs Baseline | 6.5413 [1.1144 to 11.9681] | 0.9244 [-6.7736 to 8.6224]
  Week 18 vs Baseline | 1.4568 [-4.4994 to 7.4129] | 1.1470 [-7.3990 to 9.6929]

12. Secondary Outcome: Change From Baseline in the SCORing Atopic Dermatitis (SCORAD) Score in Treated Population Compared to Placebo Population to Weeks 4, 8, 12, 16, 18.
Description: The SCORing Atopic Dermatitis (SCORAD) grading system was developed by the European Task Force on Atopic Dermatitis and has been a standard tool to assess atopic dermatitis (AD) severity in clinical studies. Six items (erythema, edema/papulation, oozing/crusts, excoriation, lichenification, and dryness) will be selected to evaluate the AD severity. The intensity of each item is graded using a 4-point scale:
  * 0 = No symptoms
  * 1 = Mild
  * 2 = Moderate
  * 3 = Severe The overall body surface area (BSA) affected by AD is evaluated (from 0 to 100%) and included in the SCORAD scores. Loss of sleep and pruritus will be evaluated by patients on a visual analog scale (0-10).
Time Frame: 18 Weeks
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 102 | 99
score on a scale
  Week 4 vs Baseline | 15.7003 [8.8854 to 22.5153] | -0.9182 [-10.6319 to 8.7955]
  Week 8 vs Baseline | 12.6334 [5.4389 to 19.8279] | -0.0799 [-10.3366 to 10.1769]
  Week 12 vs Baseline | 4.0487 [-3.5504 to 11.6478] | 5.2956 [-5.5928 to 16.1840]
  Week 16 vs Baseline | 7.3626 [0.6168 to 14.1084] | 1.8419 [-7.6580 to 11.3419]
  Week 18 vs Baseline | 1.8556 [-5.5327 to 9.2439] | 4.3232 [-6.2245 to 14.8709]

13. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs).
Description: Incidence of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) in Safety Analysis Set.
Time Frame: 20 Weeks
Population: Safety Analysis set consists of all patients who received at least one dose of the medication. SAS was the analysis population for all safety endpoints. Analysis was done according to the actual treatment patients received.
Measure: Number; unit: Adverse Events
Arm/Group | Placebo | DS107 2000mg
Number analyzed (Participants) | 110 | 109
Adverse Events
  All AEs | 58 | 62
  Serious AEs | 5 | 5
  AEs with relationship to study medication | 23 | 42
  AEs leading to death | 0 | 0
  AEs that led to withdrawal | 12 | 17

ADVERSE EVENTS:
Time Frame: Up to 20 weeks.
Description: An adverse event is any undesirable experience occurring to a patient that has signed the ICF and who has taken their first dose of the study drug, whether or not considered related to the investigational IMP(s). All Adverse Events (AEs) must be recorded in the CRF, defining relationship to IMP and severity. AEs should also be recorded by the Investigator in the patient file/notes.
Arm/Group | Placebo | DS107 2000mg
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/109
Serious Adverse Events (participants affected / at risk) | 5/110 | 5/109
Other Adverse Events (participants affected / at risk) | 53/110 | 57/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=110) | DS107 2000mg (N=109)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Coronavirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 1 (1)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=110) | DS107 2000mg (N=109)
Diarrhoea (Gastrointestinal disorders) | 4 | 21
Nausea (Gastrointestinal disorders) | 2 | 6
Headache (Nervous system disorders) | 10 | 3
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 26 | 13
Anemia (Blood and lymphatic system disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 2 | 1
Eczema Eyelids (Eye disorders) | 1 | 0
Eye Pain (Eye disorders) | 1 | 0
Macular Oedema (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sluggishness (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Breast abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Nasal herpes (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 3
Oral herpes (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pulpitis dental (Infections and infestations) | 1 | 0
Pyoderma (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Superinfection bacterial (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Tooth injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 3
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 3 | 1
White blood cell count increased (Investigations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Hypoesthesia (Nervous system disorders) | 1 | 0
Emotional distress (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Sleep disorder (Psychiatric disorders) | 2 | 1
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 | 0
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1
Erythrodermic atopic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The decision to terminate the study prematurely was based on the results from an interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03817190/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT03817190/SAP_001.pdf